CLINICAL TRIAL: NCT04427514
Title: Investigation of the Applicability of a Home Peritoneal Dialysis (CAPD= Continuous Ambulatory Peritonealis Dialysis) Application System
Brief Title: Continuous Ambulatory Peritoneal Dialysis With Telemedicine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Szeged University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: TMED_CAPD_001
Record Dates: First submitted 2020-05-19; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Peritoneal Dialysis, Continuous Ambulatory
Keywords: telemedicine
MeSH Terms: interventions — Peritoneal Dialysis, Continuous Ambulatory

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAPD group (Experimental): Standard CAPD therapy wtih telemedicine system
  Interventions: Device: Telemedicine software for data transmission and analysis in CAPD.

INTERVENTIONS:
Device: Telemedicine software for data transmission and analysis in CAPD. — Telemedicine software is related to peritoneal dialysis. With the help of a tablet device running an Android system on patients and the care team and the smart devices attached to it (scales, blood pressure monitor), patients perform measurements in their homes in connection with solution changes. The resulting data is transmitted through the telemedicine system to the care team, which can take immediate intervention if necessary and notify the patient of any change in therapy.

SUMMARY:
This clinical trial is an open-label, prospective, single-arm, single center study.

In this study is planned to involve 12 patients, who need continuous ambulatory peritonealis dialysis (CAPD). Telemedicine software is related to peritoneal dialysis. With the help of a tablet device running an Android system on patients and the care team and the smart devices attached to it (scales, blood pressure monitor), patients perform measurements in their homes in connection with solution changes. The resulting data is transmitted through the telemedicine system to the care team, which can take immediate intervention if necessary and notify the patient of any change in therapy.

DETAILED DESCRIPTION:
After enrollment, the patient is educated about the using of telemedicine system and then the standard CAPD will be continued in their home treatment supplemented with a telemedicine system.

There is a monthly follow-up visit in the CAPD therapy. Before each control visit a telemedicine doctor, for whom are available telemedicine data, decides whether a control visit is necessary. After that line the patient will be subjected to a personal check - up visit by another specialist, for whom the result of the telemedicine visit is unknown. At the end of the control visit, the doctor declares whether it could have been triggered the examination with the review of telemedicine data.

In the end of the study will be summarized the average number of visits that can be omitted and will be analyzed the extent to which the two medical opinions and the necessity of the visit matched.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years;
* Signed Informed consent form;
* Patients treated with CAPD;
* The subject communicates well with the investigator and is able to help understand and adhere to the requirements of the study plan.

Exclusion Criteria:

* The consent was withdrawn by the volunteers at any time after the information and the signed informed consent form;
* Poor general condition;
* Any disease which, in the opinion of the investigator, endangers the health of the volunteer and / or contraindicates the conduct of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
The average number of visits that can be omitted | 13 months
  In the end of the study will be summarized the average number of visits that can be omitted, and will be analyzed the extent to which the two medical opinions and the necessity of the visit matched.

CONTACTS AND LOCATIONS:
Overall Officials: Zoltán Ondrik, MD, Principal Investigator — University of Szeged, First Department of Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nakamoto H, Kawamoto A, Tanabe Y, Nakagawa Y, Nishida E, Akiba T, Suzuki H. Telemedicine system using a cellular telephone for continuous ambulatory peritoneal dialysis patients. Adv Perit Dial. 2003;19:124-9. PMID 14763048
- [Background] Li J, Wang H, Xie H, Mei G, Cai W, Ye J, Zhang J, Ye G, Zhai H. Effects of post-discharge nurse-led telephone supportive care for patients with chronic kidney disease undergoing peritoneal dialysis in China: a randomized controlled trial. Perit Dial Int. 2014 May;34(3):278-88. doi: 10.3747/pdi.2012.00268. Epub 2014 Jan 2. PMID 24385331
- [Background] Krishna VN, Managadi K, Smith M, Wallace E. Telehealth in the Delivery of Home Dialysis Care: Catching up With Technology. Adv Chronic Kidney Dis. 2017 Jan;24(1):12-16. doi: 10.1053/j.ackd.2016.11.014. PMID 28224937
- [Background] Rygh E, Arild E, Johnsen E, Rumpsfeld M. Choosing to live with home dialysis-patients' experiences and potential for telemedicine support: a qualitative study. BMC Nephrol. 2012 Mar 19;13:13. doi: 10.1186/1471-2369-13-13. PMID 22429705